CLINICAL TRIAL: NCT05752344
Title: Interstitial Cystitis: Monitoring of the Psychic State and Counseling Intervention in the COVID-19 Era
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mazza Marianna, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3499
Record Dates: First submitted 2023-02-26; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Cystitis, Interstitial
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Counseling — Professional Counseling is an activity that aims to improve the client's quality of life. Supporting his strengths and his ability to self-determination, Counseling offers a space for listening and reflection in which to explore difficulties, related to evolutionary processes, transition phase, states of crisis and reinforcement of the ability to choose or change.

SUMMARY:
The target population of this observational study is made up of all patients belonging to the Interstitial Cystitis pathway of the Gemelli University Hospital Foundation - IRCCS, who have accepted to be subjected to remote monitoring and diagnostic investigation. The aim of the study is the evaluation of some outcome parameters at the time of enrollment (T0), and at the end (T1) of subjects affected by Intersitial Cystitis who have carried out a monitoring of the dimensions of the psychic sphere concerning: depression, trait anxiety, state anxiety , well-being, self-efficacy, resilience.The objective is also to evaluate the presence of evolutionary and maturational trends in the mental set-up of the people who participated in the individual counseling intervention.

ELIGIBILITY:
Inclusion Criteria:

* Recruited subjects have a diagnosis of Interstitial Cystitis and are 18 years of age or older.

Exclusion Criteria:

* Previous or current intellectual disability in accordance with the Diagnostic and Statistical Manual of Mental Disorders, DSM-5.
* Patients who are unable to express consent and who do not have a caregiver who can give it for them.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population of this observational study is made up of all patients belonging to the Interstitial Cystitis pathway of the Gemelli University Hospital Foundation - IRCCS, who will accept to be subjected to remote monitoring and diagnostic investigation as per the proposed scheme.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSCG) | 12 months
  Administration of psychometric scales
Hospital Anxiety and Depression Scale (HADS) | 12 months
  Administration of psychometric scales

SECONDARY OUTCOMES:
Psychological General Well-Being Index (PGWBI) | 12 months
  Administration of psychometric scales

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, ROMA, Italy

IPD SHARING:
Plan to Share IPD: No